CLINICAL TRIAL: NCT04341389
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial to Evaluate the Safety and Immunogenicity of the Recombinant Novel Coronavirus Vaccine (Adenovirus Vector) in Healthy Adults Aged Above 18 Years
Brief Title: A Phase II Clinical Trial to Evaluate the Recombinant Vaccine for COVID-19 (Adenovirus Vector)
Acronym: CTII-nCoV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Biotechnology, Academy of Military Medical Sciences, PLA of China (Other)
Collaborators: CanSino Biologics Inc. (Industry); Jiangsu Province Centers for Disease Control and Prevention (Network); Hubei Provincial Center for Disease Control and Prevention (Other); Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: JSVCT089
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: COVID-19 vaccine; Ad5-nCoV; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Ad5-nCoV vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Active Comparator): 1×10^11vp of Ad5-nCoV administered through 1.0 mL intramuscular injection in the deltoid muscle on Day 0
  Interventions: Biological: Recombinant novel coronavirus vaccine (Adenovirus type 5 vector)
- Arm 2 (Active Comparator): 5×10^10vp of Ad5-nCoV administered through 1.0 mL intramuscular injection in the deltoid muscle on Day 0
  Interventions: Biological: Recombinant novel coronavirus vaccine (Adenovirus type 5 vector)
- Arm 3 (Placebo Comparator): Placebo administered through 1.0 mL intramuscular injection in the deltoid muscle on Day 0
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Recombinant novel coronavirus vaccine (Adenovirus type 5 vector) — Intramuscular injection
  Other Names: Ad5-nCoV
  Arms: Arm 1; Arm 2
Other: Placebo — Intramuscular injection
  Other Names: Control
  Arms: Arm 3

SUMMARY:
This is a phase II, randomised, double-blinded and placebo-controlled clinical trial in healthy adults above 18 years of age. This clinical trial is designed to evaluate the immunogenicity and safety of Ad5-nCoV which encodes for a full-length spike (S) protein of SARS-CoV-2.

DETAILED DESCRIPTION:
This is a phase II, randomised, double-blinded and placebo-controlled clinical trial in healthy adults above 18 years of age,inclusive, who meet all eligibility criteria. This clinical trial is designed to evaluate the immunogenicity and safety of Ad5-nCoV which encodes for a full-length spike (S) protein of SARS-CoV-2. 500 subjects will be enrolled, 250 subjects in middle-dose vaccine group, 125 subjects in low-dose and placebo group, respectively. Immunogenicity will be tested on days 0, 14, 28 and 6 months after vaccination

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years.
* Able to understand the content of informed consent and willing to sign the informed consent
* Able and willing to complete all the secluded study process during the whole 6 months study follow-up period.
* Negative in HIV diagnostic test.
* Negative in serum antibodies (IgG and IgM) screening of COVID-19.
* Axillary temperature ≤37.0°C.
* The BMI index is 18.5-30.0.
* General good health as established by medical history and physical examination.

Exclusion Criteria:

* Family history of seizure, epilepsy, brain or mental disease
* Subject allergic to any component of the investigational vaccine, or a more severe allergic reaction and history of allergies in the past.
* Woman who is pregnant, breast-feeding or positive in β-HCG (human chorionic gonadotropin) pregnancy test (urine) on day of enrollment, or become pregnant during the next 6 months
* Any acute fever disease or infections.
* History of SARS
* Major congenital defects or not well-controlled chronic illness, such as asthma, diabetes, or thyroid disease.
* Serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension without controllable drugs, etc.
* Hereditary angioneurotic edema or acquired angioneurotic edema
* Urticaria in last one year
* No spleen or functional spleen.
* Platelet disorder or other bleeding disorder may cause injection contraindication
* Faint at the sight of needles.
* Prior administration of immunodepressant or corticosteroids, antianaphylaxis treatment, cytotoxic treatment in last 6 months.
* Prior administration of blood products in last 4 months
* Prior administration of other research medicines in last 1 month
* Prior administration of attenuated vaccine in last 1 month
* Prior administration of inactivated vaccine in last 14 days
* Current anti-tuberculosis prophylaxis or therapy
* According to the judgement of investigator,various medical, psychological, social or other conditions, those could affect the subjects to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2020-04-12 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse reactions | 0-14 days post vaccination
Anti SARS-CoV-2 S IgG antibody response(ELISA) | 28 days post vaccination
Neutralizing antibody response to SARS-CoV-2 | 28 days post vaccination

SECONDARY OUTCOMES:
Occurrence of adverse events | 0-28 days post vaccination
Occurrence of serious adverse reaction | 0-6 months post vaccination
Anti SARS-CoV-2 S IgG antibody response(ELISA) | 0, 14 days and 6 months post vaccination
Neutralizing antibody response to SARS-CoV-2 | 0 and 6 months post vaccination
Neutralizing antibody response to Ad5-vector | 0, 28 days and 6 months post vaccination
IFN-γ ELISpot responses to SARS-CoV-2 spike protein | 0 and 28 days post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, MD, Principal Investigator — Jiangsu Province Centers of Disease Control and Prevention
Locations (1):
- Hubei Provincial Center for Disease Control and Prevention, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feng JL, Wang WJ, Jin PF, Zheng H, Jin LR, Xia X, Zhang XY, Li ZP, Li JX, Zhu FC. Comparison of antibody persistency through one year between one-dose and two-dose regimens of Ad5-nCoV vaccine for COVID-19. Hum Vaccin Immunother. 2023 Aug 1;19(2):2230760. doi: 10.1080/21645515.2023.2230760. PMID 37428653
- [Derived] Zhu FC, Guan XH, Li YH, Huang JY, Jiang T, Hou LH, Li JX, Yang BF, Wang L, Wang WJ, Wu SP, Wang Z, Wu XH, Xu JJ, Zhang Z, Jia SY, Wang BS, Hu Y, Liu JJ, Zhang J, Qian XA, Li Q, Pan HX, Jiang HD, Deng P, Gou JB, Wang XW, Wang XH, Chen W. Immunogenicity and safety of a recombinant adenovirus type-5-vectored COVID-19 vaccine in healthy adults aged 18 years or older: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2020 Aug 15;396(10249):479-488. doi: 10.1016/S0140-6736(20)31605-6. Epub 2020 Jul 20. PMID 32702299